CLINICAL TRIAL: NCT04286360
Title: Hematological Anomalies in Children With Rasopathy
Acronym: RAS-HEMATO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K171010J
Record Dates: First submitted 2020-01-17; First posted 2020-02-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: RAS Mutation
Keywords: RASopathie

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During childhood, patients with RASopathies (Noonan syndrome and related diseases) can harbor various hematological anomalies ranging from isolated monocytosis, myelemia, thrombocytopenia or splenomegaly to myeloproliferative disorders. These anomalies may spontaneously disappear or persist, sometimes leading to juvenile myelomonocytic leukemia. Guidelines for initial screening and subsequent hematological follow-up have recently been published in France: peripheral blood analysis should be performed in all newly diagnosed patients and followed by biannual peripheral blood analysis in infants until the age of 2 years.

In order to describe the characteristics of these abnormalities in terms of their incidence, age of occurrence, evolution and relation to genotype, we are conducting a longitudinal prospective study whose aim is to analyze peripheral blood cell counts and smears at diagnosis and one year later. In patients <3 years of age recruited at certain centers, biobanking of mononuclear cells will be performed. These data could yield a new insight into hematological anomalies in patients with RASopathies and thereby help physicians to determine the appropriate rhythm for hematological follow-up according to genotype.

ELIGIBILITY:
Inclusion Criteria:

* Age < 16 years
* Patient newly diagnosed with genetically confirmed rasopathy : Noonan syndrome, type 1 neurofibromatosis, Noonan syndrome with multiple lentigines, CBL syndrome, Costello syndrome, cardiofaciocutaneous syndrome or Legius syndrome i.e. with a germline mutation of one of these genes: PTPN11, SOS1, NRAS, RAF1, BRAF, SHOC2, MEK1, MEK2, CBL, NF1, SPRED1, KRAS, HRAS, NF1, SHOC2, LZTR1, SOS2, RIT1, RASA2, RRAS, PPP1CB, or a new gene of interest published during the recruitment period
* No history of hematological malignancy
* Written informed consent obtained from the parents
* Health insurance

Exclusion Criteria:

* History of malignant hematological pathology

Max Age: 15 Years | Sex: All
Age Groups: Child
Study Population: Patients aged 15 years old and younger with RASopathies (Noonan syndrome and related diseases)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with hematological abnormalities | at inclusion (within 6 months after diagnosis)

SECONDARY OUTCOMES:
Proportion of patients with hematological abnormalities according to genetic abnormality | at inclusion (within 6 months after diagnosis)
Proportion of patients with hematological abnormalities according to age | at inclusion (within 6 months after diagnosis)
Proportion of patients with hematological abnormalities | at 1 year after inclusion
Proportion of patients with hematological abnormalities according to age | at 1 year after inclusion
Proportion of patients with hematological abnormalities according to genetic abnormalities | at 1 year after inclusion
Evolution of proportion of patients with hematological abnormalities during childhood | at 5 years post-inclusion
Event-free survival | at one year post-inclusion
Event-free survival | at 5 years post-inclusion

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU Caen, Caen
  - CHU Lille, Lille
  - CHU Lyon, Lyon
  - CHU Marseille - Hôpital de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Necker APHP, Paris
  - Hôpital Robert Debré APHP, Paris
  - Hôpital Trousseau APHP, Paris
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided